CLINICAL TRIAL: NCT04971512
Title: A Phase 1a/1b Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of EDP-721 in Healthy Subjects (Part 1) and the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of EDP-721 in Combination With EDP-514 in Patients With Chronic Hepatitis B Virus Infection (Part 2)
Brief Title: A 2 PART STUDY EVALUATING EDP-721 IN HEALTHY SUBJECTS AND EDP-721 IN COMBINATION WITH EDP-514 IN PATIENTS WITH CHRONIC HEPATITIS B VIRUS INFECTION.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to adverse safety signals in Part 1 (HV)
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: EDP 721-001
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Chronic Hepatitis B Virus Infection
Keywords: First-in-Human; Single Ascending Dose; Multiple Ascending Dose; Hepatitis B virus; HBV
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- EDP-721 HV SAD Cohorts (Experimental): EDP-721 Dose 1, Dose 2, Dose 3 and Dose 4, in one single administration
  Interventions: Drug: EDP-721
- EDP-721 HV MAD Cohorts (Experimental): EDP-721 Dose 1, Dose 2 and Dose 3, once daily for 14 days
  Interventions: Drug: EDP-721
- EDP-721 HV SAD Placebo Cohort (Placebo Comparator): Matching placebo, in one single administration
  Interventions: Drug: Placebo (Part 1)
- EDP-721 HV MAD Placebo Cohort (Placebo Comparator): Matching placebo, once daily for 14 days
  Interventions: Drug: Placebo (Part 1)
- EDP-721+ EDP-514 HBV MAD Cohorts (Experimental): EDP-721 once daily for 14 days followed by EDP-721+EDP-514 once daily for 28 days
  Interventions: Drug: EDP-721 (Part 2); Drug: EDP-514
- EDP-721+ EDP-514 HBV MAD Placebo Cohorts (Placebo Comparator): Matching placebo once daily for 42 days
  Interventions: Drug: Placebo (Part 2)

INTERVENTIONS:
Drug: EDP-721 — Oral administration (Part 1)
  Arms: EDP-721 HV MAD Cohorts; EDP-721 HV SAD Cohorts
Drug: Placebo (Part 1) — Placebo to match EDP-721, oral administration (Part 1)
  Arms: EDP-721 HV MAD Placebo Cohort; EDP-721 HV SAD Placebo Cohort
Drug: EDP-721 (Part 2) — Oral administration (Part 2)
  Arms: EDP-721+ EDP-514 HBV MAD Cohorts
Drug: Placebo (Part 2) — Placebo to match EDP-721 (Part 2)
  Arms: EDP-721+ EDP-514 HBV MAD Placebo Cohorts
Drug: EDP-514 — Oral administration
  Arms: EDP-721+ EDP-514 HBV MAD Cohorts
Drug: Placebo (Part 2) — Placebo to match EDP-514
  Arms: EDP-721+ EDP-514 HBV MAD Placebo Cohorts

SUMMARY:
Part 1 is a randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, and pharmacokinetics of single and multiple ascending doses of EDP-721 in healthy subjects.

Part 2 is a randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics and antiviral activity of EDP-721 in combination with EDP-514 in patients with chronic hepatitis B virus infection.

ELIGIBILITY:
Part 1 (HV Population):

Inclusion Criteria:

* An informed consent document signed and dated by the subject.
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 65 years, inclusive.

Exclusion Criteria:

* Clinically relevant evidence or history of illness or disease.
* Pregnant or nursing females.
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection.
* A positive urine drug screen at screening or Day -1.
* Current tobacco smokers or use of tobacco within 3 months prior to screening.
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy).
* History of regular alcohol consumption.
* Receipt of any vaccine, an investigational agent or biological product within 28 days or 5 times the t½, whichever one is longer, prior to first dose.

Part 2 (CHB Population)

Inclusion Criteria (Nuc-Suppressed CHB Population)

* An informed consent document signed and dated by the subject.
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 70 years, inclusive
* HBsAg detectable in serum/plasma at Screening and in the most recent HBsAg serum/plasma testing at least 6 months previously.
* HBV DNA levels:

  * A Screening HBV DNA level in serum/plasma that is <LLOQ and
  * No HBV DNA serum/plasma test values ≥LLOQ over the previous 12 months (using an approved test)
* CHB subjects must have been on their prescribed HBV NUC treatment with no change in regimen for 12 months prior to Screening

Inclusion Criteria (Viremic CHB Population):

* An informed consent document signed and dated by the subject.
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 70 years, inclusive
* HBsAg detectable in serum/plasma at Screening and in the most recent HBsAg serum/plasma testing at least 6 months previously.
* HBV DNA levels:

  * For subjects who are HBeAg positive at Screening, a Screening HBV DNA level in serum/plasma that is ≥20,000 IU/ml, or
  * For subjects who are HBeAg negative at Screening, a Screening HBV DNA level in serum/plasma that is ≥2,000 IU/mL, and
  * For all subjects, no HBV DNA serum/plasma test values <1,000 IU/ml over the previous 12 months (using an approved test)
* CHB subjects must not have been on prescribed anti-HBV treatment, specifically pegIFN and/or NUC therapy for at least 12 months prior to Screening

Exclusion Criteria (Nuc-Suppressed and Viremic CHB Population):

* A documented prior diagnosis of cirrhosis
* Pregnant or nursing females
* Coinfection with human immunodeficiency virus (HIV), HCV, HDV, HAV, or HEV
* Chronic liver disease of a non-HBV etiology; coexisting liver or biliary diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Safety measured by adverse events | Up to 8 Days in HV SAD Cohorts
Safety measured by adverse events | Up to 21 Days in HV MAD Cohorts
Safety measured by adverse events | Up to 70 Days in NUC-suppressed CHB MAD Cohorts
Safety measured by adverse events | Up to 98 Days in Viremic CHB MAD Cohorts

SECONDARY OUTCOMES:
Cmax of EDP-721 | Up to 6 Days in HV SAD Cohorts
AUC of EDP-721 | Up to 6 Days in HV SAD Cohorts
Cmax of EDP-721 | Up to 18 Days in HV MAD Cohorts
AUC of EDP-721 | Up to 18 Days in HV MAD Cohorts
Cmax of EDP-721 alone and in combination with EDP-514 | Up to 28 Days in All CHB MAD Cohorts
AUC of EDP-721 alone and in combination with EDP-514 | Up to 28 Days in All CHB MAD Cohorts
Cmax of EDP-514 in combination with EDP-721 | Up to 28 Days in All CHB MAD Cohorts
AUC of EDP-514 in combination with EDP-721 | Up to 28 Days in All CHB MAD Cohorts
Change from baseline in HBV DNA Viral Load Assay | Through Day 28 in All CHB MAD Cohorts
Change from baseline in quantitative HBsAg | Through Day 28 in All CHB MAD Cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- New Zealand Clinical Research Ltd, Auckland, New Zealand